CLINICAL TRIAL: NCT06547788
Title: LEFT ATRIAL MONITORING IN PATIENTS BEFORE AND AFTER MITRAL SURGERY - LAMBDA STUDY
Acronym: LAMBDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240059
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease; Heart Failure
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitral valve repair with creation of an 8m inter-atrial shunt (Experimental)
  Interventions: Other: Mitral valve repair with creation of an 8 mm inter-atrial shunt
- Mitral valve repair without a shunt (Active Comparator)
  Interventions: Other: Mitral valve repair with creation of an 8 mm inter-atrial shunt

INTERVENTIONS:
Other: Mitral valve repair with creation of an 8 mm inter-atrial shunt — Mitral valve repair with creation of an 8 mm inter-atrial shunt

SUMMARY:
Mitral valve leakage, or mitral regurgitation (MR), is associated with heart failure symptoms including shortness of breath, fatigue, irregular heart rate. When left untreated, it may cause death. Patients with MR can be divided in two broad groups: those with primary MR, caused by disease of the mitral valve structures, and those with secondary MR, due to dilation of the heart chambers. Our study focuses on patients with primary MR.

The standard treatment for severe symptomatic primary MR is mitral valve surgery, a type of open-heart surgery. The outcomes following this procedure are excellent, however, a subset of patients continue to experience heart failure symptoms after surgery due to very high pressures in the heart, more specifically in the left atrium, which is one of the four heart chambers. This is called functional mitral stenosis (FMS).

Previous studies have shown that creating a small opening between the left and right atria can help relieve the pressure inside the left atrium. We would like to determine whether creating this opening between the two atria at the time of mitral valve surgery can help prevent FMS. To answer this question, we will study two groups of patients who need mitral valve surgery for primary MR. The first group will undergo mitral valve surgery, along with the creation of the opening between the two atria. The second group will undergo mitral valve surgery alone. We will then compare the outcomes between both groups, namely with regards to their heart failure symptoms after open-heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Severe (4+) symptomatic Carpentier Type II MR due to degenerative disease
* Planned surgical mitral valve repair
* Right-to-left atrial pressure gradient ≥ 5 mmHg at baseline
* Pulmonary vascular resistance ≤ 4 Wood units

Exclusion Criteria:

* Secondary causes of MR and mixed mitral valve disease
* Infective endocarditis within 30-days
* Any prior mitral valve intervention
* Need for emergency intervention or surgery
* Left ventricular ejection fraction 2+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: recruitment rate | 30 Months
  Process, Resources, Management, Scientific
Feasibility: Success rate of intervention | 30 Months
  Process, Resources, Management, Scientific
Feasibility: Study follow-up rate and length | 30 Months
  Process, Resources, Management, Scientific

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, Dr., Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No